CLINICAL TRIAL: NCT03244189
Title: Prevention of Urinary Stones With Hydration
Acronym: PUSH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00083271; 1U01DK110988 (NIH)
Record Dates: First submitted 2017-08-02; First posted 2017-08-09 (Actual); Results first posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Urinary Stones
Keywords: Urinary Stone Disease; Kidney Stone; Urinary Calculi
MeSH Terms: conditions — Urinary Calculi; Kidney Calculi

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The Principal Investigator and site investigators, along with the primary study statistician will remind blinded throughout the trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants in the intervention arm will receive an individualized "fluid prescription", which will be the additional volume of fluid intake needed to maintain a study-specified urine output. This fluid will be consumed from and measured by a smart water bottle. The intervention arm also includes a behavioral program that consists of financial incentives and structured problem solving (SPS) to maintain the recommended fluid intake.
  Interventions: Behavioral: Fluid prescription; Behavioral: Financial incentive; Behavioral: Structured Problem Solving
- Control (No Intervention): Participants in the control arm will receive standard care instructions according to American Urological Association (AUA) guidelines to increase overall fluid consumption to achieve study-specified urine output. They will also receive a "smart" water bottle with capability to self-monitor their fluid intake.

INTERVENTIONS:
Behavioral: Fluid prescription — The additional amount of fluid that the participant will need to consume each day, using the smart water bottle, in order to meet the study-specified urine output. This fluid is in addition to any other sources of fluid (ex. cups of coffee, bottled sports drink) that the participant consumes each day.
  Arms: Intervention
Behavioral: Financial incentive — Participants in the Intervention Arm who meet their fluid intake goal on randomly selected days will receive a small payment for that day.
  Arms: Intervention
Behavioral: Structured Problem Solving — Structure Problem Solving involves interactions with health coaches to help participants develop feasible solutions to overcoming personal barriers to maintaining the prescribed fluid intake.
  Arms: Intervention

SUMMARY:
A randomized clinical trial to investigate the impact of increased fluid intake and increased urine output on the recurrence rate of urinary stone disease (USD) in adults and children. The primary aim of the trial is to determine whether a multi-component program of behavioral interventions to increase fluid intake will result in reduced risk of stone disease progression over a 2-year period.

DETAILED DESCRIPTION:
This is a two arm randomized controlled trial that incorporates pragmatic features, an adaptable intervention, patient choice, and remote monitoring of fluid intake through a "smart" water bottle. The study period is 24 months and will enroll approximately 1642 participants. Randomization will be stratified within a study site by age (adult vs. adolescent) and first time vs. recurrent stone former.

Intervention and control arm study participants will receive a smart water bottle that records daily fluid consumption, usual care including guideline-based recommendations of adequate fluid intake to decrease kidney stone recurrence, and periodic 24 hour urine collections, imaging (low-dose CT scan or ultrasound) and follow-up questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 12 years
2. At least 1 symptomatic stone event (passage or procedural intervention) within 3 years prior to enrollment or a symptomatic stone event within 5 years if the patient also has new stone formation detected on imaging during the last 5 years. Symptomatic stone defined as any of the following:

   1. Stone passage
   2. Procedural intervention
   3. Radiographically or ultrasonographically confirmed stone with any of the following:

   i. Gross hematuria ii. Renal colic or atypical abdominal pain attributed to the stone, as determined by a treating provider iii. A clinical pattern of intermittent symptoms consistent with intermittent obstruction at the ureteropelvic junction, as determined by a treating provider
3. Low 24-hr urine volume

   1. ≥18 years old: <2.0 L/day
   2. <18 years old: <25 ml/Kg/day up to 2.0L/day
4. Able to provide informed consent (parental permission for children)
5. Owning and willing to use a smartphone or other device (e.g., tablet) compatible with the study-provided wireless enabled "smart" bottle

Exclusion Criteria:

1. Spinal cord injury
2. Currently undergoing active treatment for cancer except basal cell skin cancer, or patients with a history of cancer who completed their initial therapy <1 year before screening.
3. Known infectious (struvite), monogenic or other causes of stone disease for which therapies are likely to significantly alter course of stone disease

   1. Cystinuria
   2. Primary hyperoxaluria
   3. Primary xanthinuria
   4. Primary hyperparathyroidism
   5. Sarcoidosis
   6. Medullary sponge kidney
4. History or presence of hyponatremia (serum sodium <130 mmol/L) or hypo-osmolality (serum osmolality <275 mosm/kg)
5. Study participants with comorbidities that preclude high fluid intake or prior surgery precluding high fluid intake or leading to GI fluid losses

   1. History of or current Crohn's disease, ulcerative colitis, short gut syndrome (e.g. ileostomy, bowel bypass surgery to treat obesity, small bowel resection), chronic diarrhea, or GI tract ostomy.
   2. History of malabsorptive (e.g., Roux-en-Y gastric bypass) or restrictive (e.g., sleeve gastrectomy) bariatric surgery procedures
   3. Congestive heart failure

   i. NYHA class II or greater, and/or ii. Hospital admission in the past year for heart failure d. Lung disease with a home oxygen requirement e. Chronic kidney disease (eGFR <30 ml/min/1.7 m2 over a 3-month period) i. For adults (age ≥18), we will use the CKD-Epi equation which requires the measurement of serum creatinine only. ii. For children (age <18), we will use the bedside Schwartz (CKiD) formula. f. Nephrotic syndrome (>3.5 grams of protein per 24 hours) g. Cirrhosis with ascites
6. Women who are currently pregnant or planning pregnancy within 2 years.
7. Renal transplant recipient
8. Bedridden study participants (ECOG ≥ 3)
9. Uncorrected anatomical obstruction of the urinary tract
10. History of recurrent urinary tract infections (> 3 UTI/year proven by urine culture)
11. Exclusions due to medication use:

    1. Chronic use of lithium
    2. Long-term glucocorticoid use (> 7.5 mg prednisone daily for > 30 days prior to enrollment)
    3. Intake of narcotic medication on a daily basis for >30 days prior to enrollment
    4. Supplemental Vitamin C (> 1 g daily)
12. Individuals with stones that have developed after the initiation of medications that are strongly associated with USD such as carbonic anhydrase inhibitors (acetazolamide, topiramate, zonisamide), high dose vitamin C (> 1 g daily), high dose calcium supplementation (> 1,200 mg daily) AND who have discontinued or plan to discontinue these medications.
13. Individuals with stones composed of medications that may crystallize in the urine (guaifenesin, sulfonamides, triamterene, and the protease inhibitors indinavir and nelfinavir) AND who have discontinued or plan to discontinue these medications.

    Note: Individuals who are on long-term medications that increase the risk of stone disease, who cannot stop these medications due to other chronic conditions (e.g., HIV) and who may reduce their risk for stone recurrence through increased fluid intake, will be eligible to participate in the trial. Examples of these medications include:
    1. Carbonic anhydrase inhibitors (acetazolamide, topiramate, zonisamide)
    2. Medications that may crystallize in the urine (guaifenesin, sulfonamides, triamterene, and the protease inhibitors indinavir and nelfinavir).
14. Study participants <2 yrs life expectancy
15. Non-English Speakers
16. History of Syndrome of Inappropriate Antidiuretic Hormone Secretion (SIADH)
17. Anatomical urologic abnormalities including ileal conduits, horseshoe kidney, megaureter or solitary kidney.
18. Psychiatric conditions impairing compliance with the study
19. Vulnerable population (prisoner and/or cognitive impairment that the investigator feels will impact the study participant's ability to participate in the protocol)
20. Individual who will be unable to participate in the protocol in the judgment of the investigator.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1658 (Actual)
Dates: Start 2017-10-04 (Actual); Primary Completion 2024-05-18 (Actual); Study Completion 2024-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Scales, MD, MSHS, Principal Investigator — Duke University
Locations (8):
- United States (8):
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St. Louis, St Louis, Missouri
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital, Dallas, Texas
  - University of Texas Southwestern, Dallas, Texas
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Data and samples, for subjects who consent to sharing, will be sent to the NIDDK Data and Biological Samples Repository following database lock.
Supporting Information: Study Protocol, ICF, CSR, Analytic Code
Time Frame: 2 years after the last visit of the last participant randomized.
Access Criteria: Anyone with access to the NIDDK Data and Biological Samples Repository
URL: https://repository.niddk.nih.gov/home/

REFERENCES:
- [Derived] Wessells H, Lieske JC, Lai HH, Al-Khalidi HR, Desai AC, Harper JD, Kirkali Z, Maalouf NM, McCune R, Reese PP, Scales CD, Tasian GE; NIDDK Urinary Stone Disease Research Network. Adjudication of Self-reported Symptomatic Stone Recurrence in the Prevention of Urinary Stones With Hydration Trial. Urology. 2024 Dec;194:27-35. doi: 10.1016/j.urology.2024.08.026. Epub 2024 Sep 4. PMID 39242045
- [Derived] Reese PP, Shah S, Funsten E, Amaral S, Audrain-McGovern J, Koepsell K, Wessells H, Harper JD, McCune R, Scales CD Jr, Kirkali Z, Maalouf NM, Lai HH, Desai AC, Al-Khalidi HR, Tasian GE. Using structured problem solving to promote fluid consumption in the prevention of urinary stones with hydration (PUSH) trial. BMC Nephrol. 2024 May 28;25(1):183. doi: 10.1186/s12882-024-03605-y. PMID 38807063
- [Derived] Scales CD Jr, Desai AC, Harper JD, Lai HH, Maalouf NM, Reese PP, Tasian GE, Al-Khalidi HR, Kirkali Z, Wessells H; Urinary Stone Disease Research Network. Prevention of Urinary Stones With Hydration (PUSH): Design and Rationale of a Clinical Trial. Am J Kidney Dis. 2021 Jun;77(6):898-906.e1. doi: 10.1053/j.ajkd.2020.09.016. Epub 2020 Nov 16. PMID 33212205
- See also: The Urinary Stone Disease Research Network (USDRN) website. The USDRN is the program conducting the PUSH study. — http://usdrn.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention | Control
Started | 826 | 832
Completed | 676 | 691
Not Completed | 150 | 141
Not completed — Death | 0 | 2
Not completed — Lost to Follow-up | 92 | 107
Not completed — Physician Decision | 4 | 2
Not completed — Pregnancy | 7 | 5
Not completed — Protocol Violation | 0 | 2
Not completed — Withdrawal by Subject | 45 | 23
Not completed — Technical Problems | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 826 | 832 | 1658
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 45 [30 to 60] | 44 [27 to 58] | 44 [29 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 469 | 477 | 946
  Male | 357 | 355 | 712
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 46 | 56 | 102
  Not Hispanic or Latino | 761 | 757 | 1518
  Unknown or Not Reported | 19 | 19 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 3 | 3
  Asian | 22 | 25 | 47
  Native Hawaiian or Other Pacific Islander | 2 | 2 | 4
  Black or African American | 55 | 58 | 113
  White | 732 | 719 | 1451
  More than one race | 7 | 14 | 21
  Unknown or Not Reported | 8 | 11 | 19
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 826 | 832 | 1658

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Symptomatic Stone Event
Description: Having a symptomatic stone event was defined as meeting any 1 of 2 criteria - stone passage or a procedural intervention for a stone (whether the stone was causing symptoms or not).
Time Frame: Baseline through approximately 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 826 | 832
Participants | 154 | 165
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Other; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.77 to 1.20]

2. Secondary Outcome: Number of Participants With Asymptomatic Formation of New Stone
Time Frame: Up to approximately 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 826 | 832
Participants | 82 | 83
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Other; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.72 to 1.37]

3. Secondary Outcome: Number of Participants With Growth of Existing Stone by ≥ 2 mm in Any Dimension
Description: Comparison of the size of any stone on first observation versus later observations or at passage. Will be measured primarily through imaging (CT scan and ultrasound).
Time Frame: Baseline through approximately 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 826 | 832
Participants | 45 | 32
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Other; Odds Ratio (OR) = 1.44, 95% CI 2-sided [0.91 to 2.29]

4. Secondary Outcome: Number of Participants With Symptomatic Stone Recurrence, Asymptomatic Stone Formation, or Increase of Existing Stone by ≥2 mm in Any Dimension
Time Frame: Baseline through approximately 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 826 | 832
Participants | 232 | 236

5. Secondary Outcome: 24-hour Urine Total Volume
Time Frame: 6, 12, 18, and 24 months
Measure: Median (95% Confidence Interval); unit: L/day
Arm/Group | Intervention | Control
Number analyzed (Participants) | 826 | 832
L/day
  6 months | 1.81 [1.30 to 2.38] | 1.58 [1.10 to 2.18]
  12 months | 1.70 [1.24 to 2.29] | 1.57 [1.14 to 2.20]
  18 months | 1.70 [1.25 to 2.26] | 1.55 [1.13 to 2.09]
  24 months | 1.55 [1.18 to 2.10] | 1.47 [1.02 to 20.3]

6. Secondary Outcome: Costs of Study Interventions and Treatments for USD During the Follow-up Period
Description: To estimate study intervention costs, we will use a tool specifically designed to estimate costs associated with patient-centered interventions (R01NR011873). The costs of medical resource use will be assigned based on payment schedules (e.g., Medicare). To incorporate potential differences in health-related quality of life experienced by participants in the cost-effectiveness analysis, health state utilities will be estimated from existing literature. Full details of the economic analysis will be specified in the Economic Statistical Analysis Plan.
Time Frame: Baseline through approximately 24 months
Reporting Status: Not Posted, anticipated posting 2025-12

7. Secondary Outcome: Comprehensive Assessment of Self-Reported Urinary Symptoms (CASUS)
Description: The CASUS is a tool used to assess lower urinary tract symptoms (LUTS) in individuals, providing a comprehensive evaluation of various urinary issues. It's designed to capture a wide range of symptoms, including storage, voiding, post-micturition, urgency, incontinence, and abnormal bladder sensations. The total score ranges from 0 to 38, where a higher score indicates greater urinary symptoms.
Time Frame: Baseline, 6, 12, 18, and 24 months
Population: Participants with CASUS data available at each timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 658 | 661
score on a scale
  Baseline | 6.11 (3.298) | 5.94 (3.311)
  6 months: number analyzed (Participants) | 549 | 548
  6 months | 6.23 (3.197) | 6.11 (3.280)
  12 months: number analyzed (Participants) | 507 | 507
  12 months | 6.26 (3.442) | 6.05 (3.517)
  18 months: number analyzed (Participants) | 440 | 459
  18 months | 6.11 (3.267) | 6.11 (3.459)
  24 months: number analyzed (Participants) | 535 | 540
  24 months | 6.00 (3.283) | 6.01 (3.373)

ADVERSE EVENTS:
Time Frame: Up to approximately 24 months
Description: "Hyponatremia requiring hospitalization" was the only Serious Adverse Event (SAE) collected for the study. "Asymptomatic hyponatremia" was the only non-serious AE collected.
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/826 | 2/832
Serious Adverse Events (participants affected / at risk) | 0/826 | 0/832
Other Adverse Events (participants affected / at risk) | 12/826 | 2/832
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention (N=826) | Control (N=832)
Hyponatremia requiring hospitalization (Metabolism and nutrition disorders) | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention (N=826) | Control (N=832)
Asymptomatic hyponatremia (Metabolism and nutrition disorders) | 12 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-04): https://cdn.clinicaltrials.gov/large-docs/89/NCT03244189/Prot_SAP_000.pdf